CLINICAL TRIAL: NCT00855933
Title: A Controlled Clinical Study to Determine the Gingivitis Benefit of Flossing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008110
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control - no flossing (No Intervention): Subjects brushed thoroughly for one minute with Crest® Cavity Protection toothpaste and an Oral-B® Indicator soft, manual toothbrush once daily.
- Experimental Floss (Experimental): Subjects brushed thoroughly for one minute with Crest® Cavity Protection toothpaste and an Oral-B® Indicator soft, manual toothbrush once daily. Subjects flossed once daily with the experimental floss.
  Interventions: Device: Experimental Floss

INTERVENTIONS:
Device: Experimental Floss — Experimental Glide® floss with cetylpyridinium chloride (~13% dry weight CPC)
  Other Names: Glide®; floss; cetylpyridinium chloride; CPC
  Arms: Experimental Floss

SUMMARY:
This is a randomized, controlled, examiner-blind, parallel group, four week clinical study comparing brushing plus flossing to brushing alone in healthy adults with mild-to-moderate gingivitis.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* physically able to floss his/her teeth;
* refrained from performing oral hygiene the morning of the Baseline visit;
* have measurable gingivitis on at least 5 test sites;
* in good general health.

Exclusion Criteria:

* severe periodontal disease
* atypical discoloration or pigmentation in the gingival tissue;
* meaningful malocclusion of the anterior teeth;
* fixed facial orthodontic appliances;
* use of antibiotics within two weeks of the baseline visit and at any time during the study;
* any diseases or conditions that could be expected to interfere with the subject safely completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Biesbrock, DMD, PhD, Study Director — Procter and Gamble
Locations (2):
- Dr. Geza Terézhalmy, DDS , MA, San Antonio, Texas, United States
- Luis R. Archila, DDS, Guatemala City, Guatemala

RESULTS

PARTICIPANT FLOW:
Groups:
- Brushing Only: Control - Subjects will refrain from flossing. Subjects will brush teeth Crest® Cavity Protection toothpaste and Oral-B® Indicator soft, manual toothbrush once daily.
- Brushing + Flossing: Experimental - Subjects will floss once daily with the experimental floss. Subjects will brush teeth Crest® Cavity Protection toothpaste and Oral-B® Indicator soft, manual toothbrush once daily.
Period: Overall Study
Arm/Group | Brushing Only | Brushing + Flossing
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brushing Only | Brushing + Flossing | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.5 (10.08) | 27.8 (9.41) | 28.7 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Guatemala | 30 | 30 | 60
Whole Mouth Average Lobene Modified Gingival Index [Mean (Standard Deviation); unit: Units on a scale] | 2.41 (0.28) | 2.38 (0.27) | 2.40 (0.27)

OUTCOME MEASURES:

1. Primary Outcome: Whole Mouth Lobene Modified Gingival Index Between the Brushing Only Group and the Brushing + Flossing Group [30 Days] Units on the MGI Scale
Description: A whole-mouth average Lobene Modified Gingival Index was calculated by summing the scores and dividing by the number of sites graded (excludes missing teeth & sites not graded). Whole mouth average can range from 0 (normal) to 4 (severe inflammation).
  For each tooth, six gingival areas (distobuccal, buccal, mesiobuccal, mesiolingual, lingual, and distolingual) were scored using the following scale: 0=Normal (Absence of inflammation, 1=Mild inflammation (slight change in color, little change in texture) of any portion of but not the entire marginal or papillary gingival unit, 2=Mild inflammation criteria as above but involving the entire marginal or papillary gingival unit, 3=Moderate inflammation (moderate glazing, redness, edema, and/or hypertrophy) of the marginal or papillary gingival unit, 4=Severe inflammation (marked redness, edema and/or hypertrophy, spontaneous bleeding or ulceration) of the marginal or papillary gingival unit.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Brushing Only | Brushing + Flossing
Number analyzed (Participants) | 30 | 30
units on a scale | 1.84 (0.047) [-0.03 to 0.24] | 1.73 (0.047) [-0.03 to 0.24]
Statistical Analysis 1: Comparison: Brushing Only vs Brushing + Flossing; Test type: Superiority or Other; p = 0.126, ANCOVA — a priori threshold for statistical significance = 0.05; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.03 to 0.24], Standard Error of Mean 0.066 — 2-sided with the significance level set at 5%

ADVERSE EVENTS:
Arm/Group | Brushing Only | Brushing + Flossing
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days